CLINICAL TRIAL: NCT05058989
Title: The Evaluation of the Pathophysiology of Varicose Veins in Pregnancy
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 20HH5790
Record Dates: First submitted 2021-09-14; First posted 2021-09-28 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Varicose Veins; Varicose Veins of Lower Limb; Chronic Venous Insufficiency; Varicose; Vessel
Keywords: CVI; VV
MeSH Terms: conditions — Varicose Veins | interventions — Ultrasonography, Doppler, Duplex; Photoplethysmography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — There will be two blood samples that will be carried out for two types of analysis:
  1. DNA Genomic testing.
  2. Hormonal blood test (Estriol (E3) and progesterone serum).
  Each hormonal blood samples results including Estroil (E3) and progesterone serum levels will be correlated with the results of the next follow up to provide comprehensive information about increased hormonal levels in pregnancy and varicose veins development.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women who are aged between 18 to 47 years old (childbearing age).: These patients must be willing to be followed up for 1 year and agreeing to give the informed consent. Recruitment period will take up to three months. Follow up period will be conducted at the end of first, second and third trimester and three months after giving birth.
  Interventions: Diagnostic Test: Advanced ultrasound measurements (Duplex ultrasound (DUS) and Vector flow imaging (VFI); Other: Clinical interventions and procedures

INTERVENTIONS:
Diagnostic Test: Advanced ultrasound measurements (Duplex ultrasound (DUS) and Vector flow imaging (VFI) — PPG is a non-invasive method used to evaluates the severity venous reflux by measuring the venous refiling time (VRT).The principal of PPG works by using a small light source and a photoelectric cell attached to the skin in the medial supramalleolar area of the leg (the distal lower medial area of the leg).
  Other Names: photoplethysmography (PPG) technique
Other: Clinical interventions and procedures — First trimester (0-13 weeks):
  * Consent
  * Clinical data collection
  * Blood samples (genomic+ hormonal)
  * Duplex ultrasound
  * Vector flow imaging (advanced ultrasound software)
  * Truncated cone tool (measuring leg circumference using a tape measure)
  * PPG
  * AVVQ (Aberdeen varicose veins questionaire)
  Second trimester (14-26 weeks):
  * Clinical data collection
  * Blood sample (hormonal only)
  * DUS
  * VFI
  * Truncated cone tool
  * PPG
  * AVVQ
  Third trimester (27-40 weeks):
  Same as second trimester
  Three months after giving birth:
  Same as second trimester

SUMMARY:
Varicose veins (VV) are the early sign of Chronic venous insufficiency (CVI) which are characterised by abnormal tortuosity and dilatation of superficial veins of lower limb extremities. Factors for the development of VV exist in literature. However, the exact mechanism remains unclear. The prevalence of VV are greater in women compared to men and also higher in pregnant women compared to non-pregnant women which make pregnant women at higher risk of developing VV. Furthermore, complications of VV have negative impacts on patients' quality of life and health care budget. Therefore, better understanding of the cause of VV can contribute in better quality of life to the patient and provide valuable insights to help in reducing health care cost. The present study will investigate the contribution of both mechanical and chemical factors in pregnant women by taking blood samples for genomic testing, using Duplex ultrasound, vector flow imaging, limb volume assessment using Truncated cone tool, assessment of iliac vein compression using Photoplethysmography (PPG) technique, hormonal blood test and assessing patient's quality of life using Aberdeen Varicose Veins Questionnaire (AVVQ).

DETAILED DESCRIPTION:
Initially, patients will be approached by a member of the direct care team in the Maternity outpatients' departments in the following hospitals: West Middlesex hospital, Queen Charlotte's and Chelsea hospital and St Mary's hospital. This will be managed by experienced research professionals in the area of vascular surgery. If a patient is prepared to discuss their potential role in this research, then the researchers will discuss the study and recruitment details at the patient's convenience. Recruitment is completely voluntary and will not affect their routine care, this will be made clear during the discussion regarding the research, and again during the consenting process. Time will be made available for any questions and for the patient to consider recruitment in their own time. Patients will be required to consent before any study-related procedures are carried out. Then her personal identifiable data will be coded and pseudonymised.

The recruited patient will be interviewed to obtain clinical information that is essential for robust analysis. This clinical information will include standard demographic form which will be used for all patients in each follow up in order to record and gather important information which represents the composition of the target population. Gathered data will include patients' details; patients name, day of visit, hospital name, ID number, date of birth. Furthermore, this demographic form will record potential risk factors which may associate with VV development such as race, number of pregnancies, family history of venous disease, BMI which include weight and height, occupational factors, smoking, alcohol consumption and diet. Any complications arising from pregnancy will be also recorded. Finally, this proposed study will only record fetal weight in second and third trimester to correlate increased fetal weight with potential venous pathology.

First, patients will be asked to fill the demographic form then will be asked to stand on a scale to measure the weight. Height will be recorded by bringing the horizontal measure down to rest on the top of the participants head. Following this, patient will be asked to sit while measurements are recorded in a relevant source data sheet.

Next, the patient will be asked to stand on a step facing the sonographer to assess the incidence of varicose veins using Duplex ultrasound (DUS) and vector flow imaging (VFI). While patient is standing, Truncated cone tool will be performed immediately by measuring leg circumferences in each segments of each limb to produce accurate measurements of lower limbs volume. Following this, patient will be asked to sit on a chair for perform Iliac vein compression test (venous outflow function) using photoplethysmography (PPG) technique. Finally, patient's quality of life assessment will be evaluated by using Aberdeen Varicose Veins Questionnaire (AVVQ) check list. Thereafter, the patient will be thanked for their participation and excused.

Clinical Laboratory tests will be managed and performed by experienced research professionals in the area of vascular surgery. Four appointments will be arranged for each patient to investigate DNA genomic testing and Estriol (E3) and progesterone hormonal testing. First appointment during first trimester will include both genomic DNA and hormonal blood tests. The three remaining appointments in the second trimester, third trimester and three months after giving birth will include hormonal blood samples only. Patients will be entitled to exit the study at any time without providing a reason, this is clearly stated on our information sheet and consent form. Verbal consent will be requested before all follow-up ultrasound scans.

Researchers will ensure that demographic data, ultrasound data, lower limb volume and iliac vein compression measurements, histopathological results and quality of life assessment results will be collected and stored in such a way that confidentiality is preserved. All data will be pseudonyms by replacing names with research codes and by keeping any identifying information separate from the main dataset.

The data will be analysed with the help of the Imperial College statistics department. The results of this study may be presented at local, national or international meetings or submitted for publication in a peer-reviewed journal. From a patient's perspective, all data will be pseudonyms before the statistical analysis phase of the study and plans to publish the results of the study are made clear in our patient information sheet.

Data and all appropriate documentation will be stored for a minimum of 10 years after the completion of the study, including the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are willing to be followed up for 1 year and agreeing to give the informed consent will be included in the inclusion criteria.

Exclusion Criteria:

* Any incomplete cases such as intrauterine death.
* Participants who fail to attend the scans after their first visit will be excluded.
* Patients with congenital vascular abnormalities/syndromes such as Klippel Klippel-Trenaunay syndrome.
* Patients who are unable to provide consent.
* Anyone who are taking part in any other research.
* Potential participants who might not adequately understand verbal explanations or written information given in English, or who have special communication needs.

  * Patients with signs of acute deep vein thrombosis.
  * Patient suffered from severe injury of their great-saphenous vein

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women in their first trimester who are willing to be followed up for 1 year and agreeing to give the informed consent will be included in the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
The patency of the vein, the blood flow direction (antegrade/retrograde) and the peak reflux velocity are evaluated by Duplex ultrasound parameters. | 1 year, in each follow up (first, second, third trimester and three months after giving birth)
  Blood vein has to be patent to exclude blood clots, blood flow direction has to be antegrade to exclude backward flow (reflux) and peak reflux velocity has to be less than 0.5 seconds to be considered normal.

SECONDARY OUTCOMES:
The patency of the vein, the blood flow direction (antegrade/retrograde) and the peak reflux velocity are evaluated by Vector flow imaging. | 1 year, in each follow up (first, second, third trimester and three months after giving birth)
  Blood vein has to be patent to exclude blood clots, blood flow direction has to be antegrade to exclude backward flow (reflux) and peak reflux velocity has to be less than 0.5 seconds to be considered normal.
Measuring the lower limb volume by Truncated cone tool. | 1 year, in each follow up (first, second, third trimester and three months after giving birth)
  Measuring legs circumferences at two points C1 and C2 and the height between them (H) and then applying an equation.
Measuring the iliac vein compression using the PPG technique. | 1 year, in each follow up (first, second, third trimester and three months after giving birth)
  This technique measures the severity of venous reflux by measuring Venous refiling time (VRT) , (Abnormal less than 20 sec).
Genomic blood test | Through study completion, an average of 1 year.
  Using a blood sample to assess the patient DNA (to analyze genes that associate with the development of varicose veins ) and correlating these findings with the UK biobank study.
Hormonal blood test | 1 year, in each follow up (first, second, third trimester and three months after giving birth)
  Using a blood sample to assess two hormones (Estriol (E3) and progesterone serum levels.
The impact of varicose veins on the patient quality of life | 1 year, in each follow up (first, second, third trimester and three months after giving birth)
  Patient's quality of life will be measured using Aberdeen varicose vein questionaire (AVVQ).

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Aslam, PhD, Study Director — Academic Supervisor
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ismail L, Normahani P, Standfield NJ, Jaffer U. A systematic review and meta-analysis of the risk for development of varicose veins in women with a history of pregnancy. J Vasc Surg Venous Lymphat Disord. 2016 Oct;4(4):518-524.e1. doi: 10.1016/j.jvsv.2016.06.003. Epub 2016 Aug 4. PMID 27639009
- [Background] Evans CJ, Fowkes FG, Hajivassiliou CA, Harper DR, Ruckley CV. Epidemiology of varicose veins. A review. Int Angiol. 1994 Sep;13(3):263-70. PMID 7822904
- [Background] Fukaya E, Flores AM, Lindholm D, Gustafsson S, Zanetti D, Ingelsson E, Leeper NJ. Clinical and Genetic Determinants of Varicose Veins. Circulation. 2018 Dec 18;138(25):2869-2880. doi: 10.1161/CIRCULATIONAHA.118.035584. PMID 30566020

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT05058989/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT05058989/ICF_001.pdf